CLINICAL TRIAL: NCT01706978
Title: A Comparison of Two Adjunctive Treatments in Arthroscopic Cuff Repair: Soft Tissue or Bone Trephination, a Prospective Cohort Study
Brief Title: A Comparison of Two Adjunctive Treatments in Arthroscopic Cuff Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: University of Ottawa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2009042-01H
Record Dates: First submitted 2012-07-24; First posted 2012-10-15 (Estimated); Results first posted 2020-05-06 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Rotator Cuff Tear
Keywords: rotator cuff tear
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Soft Tissue Trephination (Experimental): Ten days prior to the standard rotator cuff repair, a trephination procedure will be carried out. The trephination procedure will take approximately 30 minutes to complete and will be carried out under local anesthesia. A needle will be placed through the skin over the shoulder and either into the bone or into the edge of the cuff tendon, depending on whether you are allocated to the "bone trephination" or "soft tissue trephination" groups. The needle will be used to make 6 small holes in either bone or the tendon in the shoulder in the area where the cuff is to be repaired.
  Interventions: Procedure: Soft Tissue Trephination
- Bone Trephination (Active Comparator): Ten days prior to the standard rotator cuff repair, a trephination procedure will be carried out. The trephination procedure will take approximately 30 minutes to complete and will be carried out under local anesthesia. A needle will be placed through the skin over the shoulder and either into the bone or into the edge of the cuff tendon, depending on whether you are allocated to the "bone trephination" or "soft tissue trephination" groups. The needle will be used to make 6 small holes in either bone or the tendon in the shoulder in the area where the cuff is to be repaired.
  Interventions: Procedure: Bone Trephination

INTERVENTIONS:
Procedure: Bone Trephination
  Arms: Bone Trephination
Procedure: Soft Tissue Trephination
  Arms: Soft Tissue Trephination

SUMMARY:
This Clinical Trial is being conducted to study two adjunctive treatments for rotator cuff repair; soft tissue and bone trephination. "Trephination" is a procedure that involves making small perforations either in the torn tendon near its edge, or in the bone that the tendon is repaired to. The rotator cuff is repaired by sewing the tendon down to the bone in the shoulder. Trephination is a new technique that is used in addition to the standard method of repairing the rotator cuff tendon.

This study will help to determine whether this technique improves the speed of healing, the strength and the re-tear rate of the repair. You are being asked to take part in this study because you have a tear of the rotator cuff that requires surgical treatment. A total of 90 participants will participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have failed standard non-surgical management of their rotator cuff tear, and who would benefit from a surgical repair of the cuff.
* Failed medical management will be defined as persistent pain and disability despite adequate standard non-operative management for 6 months.

Medical management will be defined as:

* The use of drugs including analgesics and non-steroidal anti-inflammatory drugs
* Physiotherapy consisting of stretching, strengthening and local modalities (ultrasound, cryotherapy, etc)
* Activity modification
* Imaging, and intra-operative findings confirming a full thickness tear of the rotator cuff.

Exclusion Criteria:

1. Characteristics of the cuff tear that render the cuff irrepairable: fatty infiltration in the muscles grade III (50%) or greater; superior subluxation of the humeral head; retraction of the cuff to the level of the glenoid rim.
2. Partial thickness cuff tears.
3. Significant shoulder comorbidities e.g. Bankart lesion, osteoarthritis
4. Previous surgery on affected shoulder e.g. Previous rotator cuff repair.
5. Patients with active worker's compensation claims
6. Active joint or systemic infection
7. Significant muscle paralysis
8. Rotator cuff tear arthropathy
9. Charcot's arthropathy
10. Significant medical comorbidity that could alter the effectiveness of the surgical intervention (eg. Cervical radiculopathy, polymyalgia rheumatica)
11. Major medical illness (life expectancy less then 1 year or unacceptably high operative risk)
12. Unable to speak or read English/French
13. Psychiatric illness that precludes informed consent
14. Unwilling to be followed for 1 year
15. Advanced physiologic age

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lapner, MD, Principal Investigator — The Ottawa Hospital; Guy Trudel, MD, Principal Investigator — University of Ottawa
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

REFERENCES:
- [Result] Campbell TM, Lapner P, Dilworth FJ, Sheikh MA, Laneuville O, Uhthoff H, Trudel G. Tendon contains more stem cells than bone at the rotator cuff repair site. J Shoulder Elbow Surg. 2019 Sep;28(9):1779-1787. doi: 10.1016/j.jse.2019.02.008. Epub 2019 Apr 26. PMID 31036422

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A number of participants who consented to be part of this study were withdrawn or excluded, prior to randomization due to study procedures not being able to be arranged pre-operatively for various reasons. A large number of participants were crossed over into another parallel study being run at The Ottawa Hospital.
Groups:
- Soft Tissue Trephination: Ten days prior to the standard rotator cuff repair, a trephination procedure will be carried out. The trephination procedure will take approximately 30 minutes to complete and will be carried out under local anesthesia. A needle will be placed through the skin over the shoulder and either into the bone or into the edge of the cuff tendon, depending on whether you are allocated to the "bone trephination" or "soft tissue trephination" groups. The needle will be used to make 6 small holes in either bone or the tendon in the shoulder in the area where the cuff is to be repaired.
  Soft Tissue Trephination
- Bone Trephination: Ten days prior to the standard rotator cuff repair, a trephination procedure will be carried out. The trephination procedure will take approximately 30 minutes to complete and will be carried out under local anesthesia. A needle will be placed through the skin over the shoulder and either into the bone or into the edge of the cuff tendon, depending on whether you are allocated to the "bone trephination" or "soft tissue trephination" groups. The needle will be used to make 6 small holes in either bone or the tendon in the shoulder in the area where the cuff is to be repaired.
  Bone Trephination
Period: Overall Study
Arm/Group | Soft Tissue Trephination | Bone Trephination
Started | 47 | 41
Completed | 38 | 35
Not Completed | 9 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Soft Tissue Trephination | Bone Trephination | Total
Number analyzed (Participants) | 47 | 41 | 88
Age, Continuous [Mean (Full Range); unit: years] | 59.5 [40 to 73] | 58.8 [42 to 75] | 59.2 [40 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 56
  Male | 19 | 13 | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 47 | 41 | 88
Hand Dominance [Count of Participants; unit: Participants]
  Non-Dominant Arm Affected | 20 | 16 | 36
  Dominant Arm Affected | 27 | 25 | 52

OUTCOME MEASURES:

1. Primary Outcome: Western Ontario Rotator Cuff Index
Description: The Western Ontario Rotator Cuff Index (WORC) is a disease specific evaluation, proven to be an accurate and valid assessment of function after shoulder replacement. The WORC is a patient-reported measure, 19-question survey. Each question is measured using a visual analog scale rated from 0-100, where higher scores mean better outcome. These scores are combined and translated into a percentage out of 100. A higher total score indicates a better outcome.
Time Frame: From baseline to up until 24-Months Post-Operative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Soft Tissue Trephination | Bone Trephination
Number analyzed (Participants) | 38 | 35
score on a scale | 82 (25) | 80 (21)

2. Secondary Outcome: American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form (ASES) Scores
Description: The ASES is a shoulder specific assessment divided into two sections: pain and activities of daily living (ADL). Pain is recorded on a visual analogue scale (0-10), lower scores indicate better outcomes. There are 10 activities of daily living questions, each are recorded on a 4 level likert scale (0-3), which a higher score indicates a better outcome. The overall score is an equal weight of the two sections and produces a score out of 100. The higher the score, the better the outcome.
Time Frame: From baseline to up until 24-Months Post-Operative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Soft Tissue Trephination | Bone Trephination
Number analyzed (Participants) | 38 | 35
score on a scale | 85 (22) | 84 (17)

3. Secondary Outcome: The Constant Score
Description: The Constant Score reflects an overall clinical functional assessment. This instrument is based on a 100-point scoring system. Subjective findings (pain, activities of daily living, and working in different positions) make up a total of 35 points. Objective measurements make up the remaining 65 points.The test is divided into four sub-categories: (1) pain is measured using 4 likert levels (15 points maximum), where a higher score indicates a better outcome; activities of daily living are measured using a likert scale, where a higher number indicates better outcomes (20 points maximum); mobility is measured by an assessor, and rated using a likert scale where a higher score indicates better outcomes (40 points maximum); finally, strength is measured by an assessor where 1 point is given per 0.5kg of force (maximum 25 points), a higher score indicates better outcomes. All categories are added together, and a total score out of 100 is given (higher score indicates better outcome).
Time Frame: From baseline to up until 24-Months Post-Operative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Soft Tissue Trephination | Bone Trephination
Number analyzed (Participants) | 38 | 35
score on a scale
  Total Score | 81 (16) | 83 (12)
  Strength | 15.9 (6.4) | 15.8 (10.3)

4. Secondary Outcome: Healing Rates
Description: Imaging parameters will be examined using ultrasound and magnetic resonance imaging (MRI). These images will be analyzed to determine healing status of the tissues post-operatively. Imaging will determine whether the tissue is healed, partially torn, or fully torn after surgery. Higher incidence of tearing will be compared between groups. A higher incidence of tearing indicates worse outcomes.
Time Frame: From surgery to up until 24-Months Post-Operative
Measure: Number; unit: percentage of participants
Arm/Group | Soft Tissue Trephination | Bone Trephination
Number analyzed (Participants) | 39 | 36
percentage of participants
  Percentage of Participants Healed | 87 | 75
  Percentage of Participants Partially-Healed | 2 | 14
  Percentage of Participants Non-Healed | 10 | 11

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the time the participant was enrolled up until 2-years post-operative for each participant.
Arm/Group | Soft Tissue Trephination | Bone Trephination
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/47 | 1/41
Other Adverse Events (participants affected / at risk) | 2/47 | 4/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Soft Tissue Trephination (N=47) | Bone Trephination (N=41)
Stroke (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Soft Tissue Trephination (N=47) | Bone Trephination (N=41)
Revision Surgery (Surgical and medical procedures) | 2 | 2
Radiating Pain into Hand (Investigations) | 0 | 1
Olecranon Fracture (Surgical and medical procedures) | 0 | 1

LIMITATIONS AND CAVEATS:
The sample size achieved would have detected a clinically significant difference based on power analysis but remains susceptible to type II error. The lack of a prospective control group also restricts the interpretation of the study finding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT01706978/Prot_SAP_000.pdf